CLINICAL TRIAL: NCT01568658
Title: Clinical and Molecular Manifestations of Neuromuscular and Neurogenetic Disorders of Childhood
Brief Title: Genetic and Physical Study of Childhood Nerve and Muscle Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120095; 12-N-0095
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-09-26

CONDITIONS: Muscular Dystrophies; Muscle Myopathies; Hereditary Spastic Paraplegias; Inherited Neuropathies; Inherited Neuromuscular Conditions
Keywords: Hereditary Myopathies; Neuropathology; Muscular Dystrophy; Natural History
MeSH Terms: conditions — Muscular Dystrophies; Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Affected probands: Affected probands over age 4 weeks and onwards with known or suspected inherited neurological disorders of childhood onset
- Healthy volunteers: Healthy volunteers will be recruited for the imaging procedures in order to establish baseline and age-range matched data on the healthy, maturing muscle, spinal cord volume and dynamic breathing
- Single patient on Idebenone: Single patient on IND expanded access of Idebenone
- Unaffected family members: Families of affected probands with known or suspected inherited neurological disorders of childhood onset

SUMMARY:
Background:

- Some nerve and muscle disorders that start early in life (before age 25), like some forms of muscular dystrophy, can run in families. However, the genetic causes of these disorders are not known. Also, doctors do not fully understand how symptoms of these disorders change over time. Researchers want to learn more about genetic nerve and muscle disorders that start in childhood by studying affected people and their family members, as well as healthy volunteers.

Objectives:

- To better understand nerve and muscle disorders that start early in life and run in families.

Eligibility:

* Individuals at least 4 weeks old with childhood-onset muscular and nerve disorders, including those who have a later onset of a disorder that typically has childhood onset.
* Affected and unaffected family members of the individuals with muscular and nerve disorders.
* Healthy volunteers at least 4 weeks old with no nerve or muscle disorders.

Design:

* Participants will be screened with a physical exam and medical history. Genetic information will be collected from blood, saliva, cheek swab, or skin samples. Urine samples may also be collected.
* Healthy volunteers and unaffected family members will have imaging studies of the muscles. These studies will include magnetic resonance imaging (MRI) and ultrasound scans. Results will be compared with those from the affected participants.
* All participants with nerve and muscle disorders will have multiple tests, including the following:
* Imaging studies of the muscles, including ultrasound and MRI scans.
* Imaging studies of the bones, such as x-rays and DEXA scans.
* Heart and lung function tests.
* Eye exams.
* Nerve and muscle electrical activity tests and biopsies.
* Video and photo image collection of affected muscles.
* Speech, language, and swallowing evaluation.
* Lumbar puncture to collect spinal fluid for study.
* Tests of movement, attention, thinking, and coordination.
* Participants with nerve and muscle disorders will return to the Clinical Center every year. They will repeat the tests and studies at these visits.

DETAILED DESCRIPTION:
Objective:

To diagnose and elucidate the underlying disease mechanism in patients with neuromuscular and neurogenetic disorders with congenital or pediatric onset (phase 1 of the protocol) and to study the natural history and mechanism of disease in neuromuscular and neurogenetic disorders of childhood (phase 2 of the protocol).

Study population:

Patients with childhood onset neuromuscular and neurogenetic disorders, their affected and unaffected family members, and healthy volunteers. Patients with later onset of a disorder that is known to typically have childhood onset will be included as well.

Design:

Diagnostic and prospective longitudinal natural history study.

Outcome Measures:

Diagnose and characterize patients with neuromuscular and neurogenetic disorders with congenital or pediatric onset and study the natural history and underlying disease mechanism. In the characterized patient population identify and develop effective outcome measures for use in future clinical trials, including applicable motor scales, quality of life scales, biomarkers from blood and urine, imaging studies, and pulmonary function tests.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Probands inclusion criteria Phase 1:

1. Aged 4 weeks and older
2. Documentation of a personal history of a childhood-onset, hereditary/familial, neurological disorder or later onset of a disease that more commonly has childhood onset. Acceptable documentation includes evaluation through any or all of the following evaluations done prior to enrollment.

   1. Medical history, including family history information
   2. Physical examination
   3. Muscle, nerve, or skin biopsy
   4. Magnetic resonance imaging (MRI)
   5. Electromyography (EMG)
   6. Nerve conduction study (NCS)
   7. Electroencephalogram (EEG)
   8. Muscle ultrasound
   9. Genetic, metabolic, or other laboratory testing such as increased serum Creatine Kinase (CK) and abnormal serum lactate/pyruvate ratio.

Exclusion criteria for probands Phase 1:

1. Individuals who are unable or unwilling to be examined
2. Minors who do not hve a parent or guardian able to provide informed consent
3. Adults seen offsite who are unable to provide their own consent

Probands inclusion criteria Phase 2:

1. Aged 4 weeks and older
2. Documentation of a defined childhood onset neuromuscular and neurogenetic disorders through phase 1 testing.

Exclusion criteria for probands Phase 2:

1. Individuals who are unable or unwilling to be examined.
2. Adults who are unable to provide their own consent and who have not previously appointed an individual with Durable Power of Attorney (DPA) or who are unable to appoint a DPA or guardian.
3. Minors who do not have a parent or guardian able to provide informed consent.
4. Adults seen offsite who are unable to provide their own consent.

Unaffected Family members - Inclusion Criteria:

1. Unaffected family members must be related by blood to a proband enrolled in the study. Biological relations may include first (parent or sibling), second (grandparents, aunts, uncles, half siblings) and third degree relatives (cousins).
2. Age 4 weeks and older.

Unaffected Family members - Exclusion Criteria:

1. Individuals whom are unable or unwilling to be examined.
2. Family members who are showing symptoms of the familial neurogenetic or neuromuscular condition (these may be enrolled as probands).
3. Neonates.
4. Adults who are unable to provide their own consent.

Healthy Volunteers - Inclusion Criteria:

1. Must be unaffected by a neurological condition.
2. Willing and able to comply with all protocol requirements and procedures, including MRI without sedation and without contrast.
3. Able to give informed assent and parent(s)/legal guardian to give informed consent in writing signed by the subject and/or parent(s)/legal guardian.

Healthy Volunteers - Exclusion Criteria:

1. Healthy volunteers who have metal objects in their body that are not MRI-safe. These include the following objects: 1) pacemakers or other implanted electrical devices; 2) brain stimulators; 3) some types of dental implants; 4) aneurysm clips (metal clips on the wall of a large artery); 5) metallic prostheses (including metal pins and rods, heart valves, and cochlear implants; 6) implanted delivery pump; 7) permanent eye liner; or 8) shrapnel fragments.
2. Healthy volunteers who have a fear of closed spaces.
3. Neonates.
4. Pregnant

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Affected probands with the following categories of childhood onset inherited neurological disorders will be enrolled:-peripheral neuropathies; -muscular dystrophies and myopathies; -congenital muscular dystrophies and congenital myopathies; -disorders of the neuromuscular junction; -motor neuron disorders; -neuromotor or movement disorders; -disorders of brain development; -neurometabolic disorders; -disorders that have a phenotype suggestive of neurogenetic or neuromuscular disease but which have not yet been genetically confirmed. Families of affected probands, with known or suspected inherited neurological disorders of childhood onset will be enrolled. Healthy volunteers will enrolled for one-time imaging procedures. A single patient with compound heterozygous FDX2 mutations will be enrolled under an emergency IND for use of Idebenone for slowing progression of subacute blindness.
Sampling Method: Non-Probability Sample
Enrollment: 9300 (Estimated)
Dates: Start 2012-03-20 (Actual)

PRIMARY OUTCOMES:
Diagnose and characterize patients with neuromuscular and neurogenetic disorders with congenital or pediatric onset and study the natural history and underlying disease mechanism. | Ongoing
In the characterized patient population identify and develop effective outcome measures for use in future clinical trials, including applicable motor scales, quality of life scales, biomarkers from blood and urine, imaging studies, and pulmonary... | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Carsten G Bonnemann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-N-0095.html